CLINICAL TRIAL: NCT00760760
Title: Impact of n-3 Polyunsaturated Fatty Acids on Adipose Tissue Inflammation in Morbidly Obese Patients
Brief Title: n-3 Polyunsaturated Fatty Acids in Obesity
Acronym: PUFA-ATI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Thomas M Stulnig, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PUFA-ATI1; OeNB12735
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Adipose Tissue Inflammation; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Omacor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- n-3 PUFA (Experimental)
  Interventions: Drug: reesterified long-chain n-3 polyunsaturated fatty acids (EPA, DHA)
- Control (Placebo Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: reesterified long-chain n-3 polyunsaturated fatty acids (EPA, DHA) — 4g daily, 8 weeks
  Other Names: Omacor®
  Arms: n-3 PUFA
Drug: control — equivalent amount of fat as butter
  Arms: Control

SUMMARY:
Inflammation in the adipose (fat) tissue is an important condition leading to metabolic derangements and cardiovascular disease in obese patients. n-3 polyunsaturated fatty acids exert anti-inflammatory effects and prevent adipose tissue inflammation in rodent obesity. This study tests the hypothesis that n-3 polyunsaturated fatty acids ameliorate adipose tissue inflammation in morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic morbidly obese patients (BMI > 40 kg/m2) supposed to undergo bariatric surgery
* Age 20-65 yrs

Exclusion Criteria:

* Acute illness within the last two week
* Known diabetes mellitus or current anti-diabetic medication
* Acquired immunodeficiency (HIV infection)
* Hepatitis or other significant liver disease
* Severe or untreated cardiovascular, renal, pulmonary disease
* Untreated or inadequately treated clinically significant thyroid disease
* Anemia
* Active malignant disease
* Inborn or acquired bleeding disorder including warfarin treatment
* Pregnancy or breast feeding
* Drug intolerability that prohibits the use of the study drug

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adipose tissue inflammation | Eight weeks of treatment

SECONDARY OUTCOMES:
Metabolic control | Eight weeks of treatment
Dependence of effects on Pparg polymorphisms | Eight weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Stulnig, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Itariu BK, Zeyda M, Leitner L, Marculescu R, Stulnig TM. Treatment with n-3 polyunsaturated fatty acids overcomes the inverse association of vitamin D deficiency with inflammation in severely obese patients: a randomized controlled trial. PLoS One. 2013;8(1):e54634. doi: 10.1371/journal.pone.0054634. Epub 2013 Jan 25. PMID 23372745
- [Derived] Itariu BK, Zeyda M, Hochbrugger EE, Neuhofer A, Prager G, Schindler K, Bohdjalian A, Mascher D, Vangala S, Schranz M, Krebs M, Bischof MG, Stulnig TM. Long-chain n-3 PUFAs reduce adipose tissue and systemic inflammation in severely obese nondiabetic patients: a randomized controlled trial. Am J Clin Nutr. 2012 Nov;96(5):1137-49. doi: 10.3945/ajcn.112.037432. Epub 2012 Oct 3. PMID 23034965